CLINICAL TRIAL: NCT05608824
Title: Evaluation of Lower Extremity Athletic Injuries and Response to Treatment Using Shear Wave Elastography and Micro-vascular Flow Imaging
Brief Title: Evaluation of Lower Extremity Athletic Injuries and Response to Treatment Using SWE and MFI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Oregon (Other)
Responsible Party: Principal Investigator, Kenton W. Gregory, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00000608
Record Dates: First submitted 2022-10-20; First posted 2022-11-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Lower Extremity Musculoskeletal Injury
Keywords: Ultrasound; Shear wave elastography; Microvascular flow imaging

STUDY DESIGN:
Masking Description: All SWE and MFI images are evaluated for quality and analyzed by qualified study physicians that are blinded to the clinical data. The analysis includes but is not limited to reading images, identifying the regions of interest, and making measurements. Clinical data will then be reviewed to validate the clinical diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Musculoskeletal injury (Experimental): Shear wave elastography and microvascular flow imaging.
  Interventions: Device: Shear wave elastography and microvascular flow imaging.

INTERVENTIONS:
Device: Shear wave elastography and microvascular flow imaging. — Subjects will undergo serial SWE and MFI imaging throughout their rehabilitation episode of care to assess changes over time, status in rehabilitation and comparison to the contralateral extremity.

SUMMARY:
Primary Objective:

To explore changes in shear wave elastography (SWE) and microvascular flow imaging (MFI) measurements from time of injury through the recovery phase of lower extremity musculoskeletal injuries to determine if a correlation exists with functional impairment.

Secondary Objective:

To develop a deep learning AI system for automated region of interest (ROI) determination for measurement of average SWE and MFI.

Methodology:

Eligible subjects with lower extremity injuries will undergo SWE and MFI measurements and complete the Lower Extremity Functional Scale questionnaire at each study visit. Clinical data related to the evaluation of the injury acquired during standard medical care of the injury will be collected from the patients' medical record such as CT or MRI scans, X-rays, physical exams and tests as well as laboratory measurements. Subjects will undergo serial SWE and MFI imaging throughout their rehabilitation episode of care to assess changes over time, status in rehabilitation and comparison to the contralateral extremity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 - 89 years;
* Able to sign an informed consent document;
* Suspected MSK injury of the lower extremity (i.e. hamstring injuries and soft tissue injuries involving the ankle).

Exclusion Criteria:

* Prior fasciotomy of same limb;
* Hemodialysis grafts of involved extremity;
* Extremity wounds preventing ultrasound imaging.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
kPa | Within 48 hours
  Tissue stiffness measured by shear wave elastography
kPa | 5 days post injury (+/- 2 days)
  Tissue stiffness measured by shear wave elastography
kPa | 6 weeks post injury (+/- 1 week)
  Tissue stiffness measured by shear wave elastography
kPa | 12 weeks post injury (+/- 1 week)
  Tissue stiffness measured by shear wave elastography
kPa | 24 weeks post injury (+/- 1 week)
  Tissue stiffness measured by shear wave elastography
Presence of blood flow | Within 48 hours
  Measured by microvascular flow imaging
Presence of blood flow | 5 days post injury (+/- 2 days)
  Measured by microvascular flow imaging
Presence of blood flow | 6 weeks post injury (+/- 1 week)
  Measured by microvascular flow imaging
Presence of blood flow | 12 weeks post injury (+/- 1 week)
  Measured by microvascular flow imaging
Presence of blood flow | 24 weeks post injury (+/- 1 week)
  Measured by microvascular flow imaging

CONTACTS AND LOCATIONS:
Overall Officials: Kenton Gregory, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - University of Oregon, Eugene, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmont PJ, Schoenfeld AJ, Goodman G. Epidemiology of combat wounds in Operation Iraqi Freedom and Operation Enduring Freedom: orthopaedic burden of disease. J Surg Orthop Adv. 2010 Spring;19(1):2-7. PMID 20370999
- [Background] Kelly JF, Ritenour AE, McLaughlin DF, Bagg KA, Apodaca AN, Mallak CT, Pearse L, Lawnick MM, Champion HR, Wade CE, Holcomb JB. Injury severity and causes of death from Operation Iraqi Freedom and Operation Enduring Freedom: 2003-2004 versus 2006. J Trauma. 2008 Feb;64(2 Suppl):S21-6; discussion S26-7. doi: 10.1097/TA.0b013e318160b9fb. PMID 18376168
- [Background] Mauser N, Gissel H, Henderson C, Hao J, Hak D, Mauffrey C. Acute lower-leg compartment syndrome. Orthopedics. 2013 Aug;36(8):619-24. doi: 10.3928/01477447-20130724-07. PMID 23937740
- [Background] Ritenour AE, Dorlac WC, Fang R, Woods T, Jenkins DH, Flaherty SF, Wade CE, Holcomb JB. Complications after fasciotomy revision and delayed compartment release in combat patients. J Trauma. 2008 Feb;64(2 Suppl):S153-61; discussion S161-2. doi: 10.1097/TA.0b013e3181607750. PMID 18376159
- [Background] Ritenour AE, Blackbourne LH, Kelly JF, McLaughlin DF, Pearse LA, Holcomb JB, Wade CE. Incidence of primary blast injury in US military overseas contingency operations: a retrospective study. Ann Surg. 2010 Jun;251(6):1140-4. doi: 10.1097/SLA.0b013e3181e01270. PMID 20485126
- [Background] Rush RM Jr, Beekley AC, Puttler EG, Kjorstad RJ. The mangled extremity. Curr Probl Surg. 2009 Nov;46(11):851-926. doi: 10.1067/j.cpsurg.2009.05.003. No abstract available. PMID 19804853
- [Background] Shadgan B, Pereira G, Menon M, Jafari S, Darlene Reid W, O'Brien PJ. Risk factors for acute compartment syndrome of the leg associated with tibial diaphyseal fractures in adults. J Orthop Traumatol. 2015 Sep;16(3):185-92. doi: 10.1007/s10195-014-0330-y. Epub 2014 Dec 28. PMID 25543232
- [Background] Kragh JF Jr, Wade CE, Baer DG, Jones JA, Walters TJ, Hsu JR, Wenke JC, Blackbourne LH, Holcomb JB. Fasciotomy rates in operations enduring freedom and iraqi freedom: association with injury severity and tourniquet use. J Orthop Trauma. 2011 Mar;25(3):134-9. doi: 10.1097/BOT.0b013e3181e52333. PMID 21321506
- [Background] McMillan TE, Gardner WT, Schmidt AH, Johnstone AJ. Diagnosing acute compartment syndrome-where have we got to? Int Orthop. 2019 Nov;43(11):2429-2435. doi: 10.1007/s00264-019-04386-y. Epub 2019 Aug 29. PMID 31468110
- [Background] Brandenburg JE, Eby SF, Song P, Zhao H, Landry BW, Kingsley-Berg S, Bamlet WR, Chen S, Sieck GC, An KN. Feasibility and reliability of quantifying passive muscle stiffness in young children by using shear wave ultrasound elastography. J Ultrasound Med. 2015 Apr;34(4):663-70. doi: 10.7863/ultra.34.4.663. PMID 25792582
- [Background] Lacourpaille L, Hug F, Bouillard K, Hogrel JY, Nordez A. Supersonic shear imaging provides a reliable measurement of resting muscle shear elastic modulus. Physiol Meas. 2012 Mar;33(3):N19-28. doi: 10.1088/0967-3334/33/3/N19. Epub 2012 Feb 28. PMID 22370174
- [Background] Nightingale KR, Palmeri ML, Nightingale RW, Trahey GE. On the feasibility of remote palpation using acoustic radiation force. J Acoust Soc Am. 2001 Jul;110(1):625-34. doi: 10.1121/1.1378344. PMID 11508987
- [Background] Ganesan S, Man CS, Lai-Fook SJ. Generation and detection of lung stress waves from the chest surface. Respir Physiol. 1997 Oct;110(1):19-32. doi: 10.1016/s0034-5687(97)00065-0. PMID 9361149
- [Background] Catheline S, Thomas JL, Wu F, Fink MA. Diffraction field of a low frequency vibrator in soft tissues using transient elastography. IEEE Trans Ultrason Ferroelectr Freq Control. 1999;46(4):1013-9. doi: 10.1109/58.775668. PMID 18238506
- [Background] Sarvazyan AP, Rudenko OV, Swanson SD, Fowlkes JB, Emelianov SY. Shear wave elasticity imaging: a new ultrasonic technology of medical diagnostics. Ultrasound Med Biol. 1998 Nov;24(9):1419-35. doi: 10.1016/s0301-5629(98)00110-0. PMID 10385964
- [Background] Bercoff J, Tanter M, Fink M. Supersonic shear imaging: a new technique for soft tissue elasticity mapping. IEEE Trans Ultrason Ferroelectr Freq Control. 2004 Apr;51(4):396-409. doi: 10.1109/tuffc.2004.1295425. PMID 15139541
- [Background] Parker KJ, Huang SR, Musulin RA, Lerner RM. Tissue response to mechanical vibrations for "sonoelasticity imaging". Ultrasound Med Biol. 1990;16(3):241-6. doi: 10.1016/0301-5629(90)90003-u. PMID 2194336
- [Background] Muthupillai R, Lomas DJ, Rossman PJ, Greenleaf JF, Manduca A, Ehman RL. Magnetic resonance elastography by direct visualization of propagating acoustic strain waves. Science. 1995 Sep 29;269(5232):1854-7. doi: 10.1126/science.7569924.
- [Background] Sarvazyan A, Hall TJ, Urban MW, Fatemi M, Aglyamov SR, Garra BS. AN OVERVIEW OF ELASTOGRAPHY - AN EMERGING BRANCH OF MEDICAL IMAGING. Curr Med Imaging Rev. 2011 Nov;7(4):255-282. doi: 10.2174/157340511798038684. PMID 22308105
- [Background] Brandenburg JE, Eby SF, Song P, Zhao H, Brault JS, Chen S, An KN. Ultrasound elastography: the new frontier in direct measurement of muscle stiffness. Arch Phys Med Rehabil. 2014 Nov;95(11):2207-19. doi: 10.1016/j.apmr.2014.07.007. Epub 2014 Jul 24. PMID 25064780
- [Background] Creze M, Nordez A, Soubeyrand M, Rocher L, Maitre X, Bellin MF. Shear wave sonoelastography of skeletal muscle: basic principles, biomechanical concepts, clinical applications, and future perspectives. Skeletal Radiol. 2018 Apr;47(4):457-471. doi: 10.1007/s00256-017-2843-y. Epub 2017 Dec 9. PMID 29224123
- [Background] Hildebrandt W, Schwarzbach H, Pardun A, Hannemann L, Bogs B, Konig AM, Mahnken AH, Hildebrandt O, Koehler U, Kinscherf R. Age-related differences in skeletal muscle microvascular response to exercise as detected by contrast-enhanced ultrasound (CEUS). PLoS One. 2017 Mar 8;12(3):e0172771. doi: 10.1371/journal.pone.0172771. eCollection 2017. PMID 28273102
- [Background] Sadeghi S, Johnson M, Bader DA, Cortes DH. The shear modulus of lower-leg muscles correlates to intramuscular pressure. J Biomech. 2019 Jan 23;83:190-196. doi: 10.1016/j.jbiomech.2018.11.045. Epub 2018 Dec 10. PMID 30563763
- [Background] Gliemann L, Mortensen SP, Hellsten Y. Methods for the determination of skeletal muscle blood flow: development, strengths and limitations. Eur J Appl Physiol. 2018 Jun;118(6):1081-1094. doi: 10.1007/s00421-018-3880-5. Epub 2018 May 14. PMID 29756164
- [Background] GREENFIELD AD, WHITNEY RJ, MOWBRAY JF. Methods for the investigation of peripheral blood flow. Br Med Bull. 1963 May;19:101-9. doi: 10.1093/oxfordjournals.bmb.a070026. No abstract available. PMID 13950177
- [Background] Jorfeldt L, Wahren J. [Leg blood supply during exercise: methodological studies with a dye dilution technic]. Nord Med. 1971 Aug 26;86(34):1009. No abstract available. Swedish. PMID 4938749
- [Background] WILD JJ, NEAL D. Use of high-frequency ultrasonic waves for detecting changes of texture in living tissues. Lancet. 1951 Mar 24;1(6656):655-7. doi: 10.1016/s0140-6736(51)92403-8. No abstract available. PMID 14814827
- [Background] Nguyen T, Davidson BP. Contrast Enhanced Ultrasound Perfusion Imaging in Skeletal Muscle. J Cardiovasc Imaging. 2019 Jul;27(3):163-177. doi: 10.4250/jcvi.2019.27.e31. Epub 2019 May 20. PMID 31161755
- [Background] Dunford EC, Au JS, Devries MC, Phillips SM, MacDonald MJ. Cardiovascular aging and the microcirculation of skeletal muscle: using contrast-enhanced ultrasound. Am J Physiol Heart Circ Physiol. 2018 Nov 1;315(5):H1194-H1199. doi: 10.1152/ajpheart.00737.2017. Epub 2018 Aug 3. PMID 30074839
- [Background] Sboros V, Tang MX. The assessment of microvascular flow and tissue perfusion using ultrasound imaging. Proc Inst Mech Eng H. 2010;224(2):273-90. doi: 10.1243/09544119JEIM621. PMID 20349819
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543